CLINICAL TRIAL: NCT00971750
Title: Comparison of Laparoscopic Ultrasound to Transabdominal Ultrasound for the Detection of Gallbladder Pathology in the Bariatric Surgical Population.
Brief Title: Laparoscopic Versus Transabdominal Ultrasound in Morbidly Obese Patients
Status: Completed | Type: Observational
Sponsor: Gundersen Lutheran Medical Foundation (Other)
Collaborators: Gundersen Lutheran Health System (Other)
Responsible Party: Principal Investigator, Kara Kallies, Advanced Research Associate, under direction of Shanu N. Kothari, MD, (PI), Gundersen Lutheran Medical Foundation
Other Study IDs: 2-03-08-009
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Results first posted 2012-07-02 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-06

CONDITIONS: Cholelithiasis; Ultrasonography; Laparoscopic Gastric Bypass
Keywords: ultrasonography; gallbladder; cholelithiasis; laparoscopic; gastric bypass; obesity; bariatric surgery
MeSH Terms: conditions — Cholelithiasis; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Ultrasound Study Group: Patients with no history of gallbladder surgery who are undergoing elective laparoscopic roux-en-Y gastric bypass that have consented to undergo a preoperative transabdominal ultrasound in addition to routine preoperative assessment for surgery.

SUMMARY:
The objective of this study is to prospectively compare laparoscopic ultrasound to transabdominal ultrasound for the detection of gallbladder pathology in obese patients presenting for laparoscopic gastric bypass. We hypothesize that laparoscopic ultrasound will be more sensitive and specific for cholelithiasis than transabdominal ultrasound in morbidly obese patients.

DETAILED DESCRIPTION:
Asymptomatic cholelithiasis is a prevalent condition in obese patients presenting for bariatric surgery. Transabdominal ultrasound (TAU) remains the gold standard for detection of cholelithiasis. The sensitivity and specificity of transabdominal ultrasound for cholelithiasis reported in literature is between 88-97% and 97-99%, respectively. The ability to detect cholelithiasis with TAU in the obese population may be inhibited due to the presence of increased subcutaneous and visceral fat. Laparoscopic ultrasound (LU) has the potential to overcome these technical challenges. In an era of minimally invasive bariatric surgery, it has been suggested that routine preoperative ultrasound TAU be performed for the detection of cholelithiasis since intraoperative palpation is not feasible. We hypothesize that laparoscopic ultrasound will be more sensitive and specific for cholelithiasis than transabdominal ultrasound in morbidly obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patients undergoing elective laparoscopic roux-en-Y gastric bypass

Exclusion Criteria:

* Prior history of gallbladder surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of patients undergoing laparoscopic gastric bypass at a community-based teaching institution.
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2003-10; Primary Completion 2010-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shanu N Kothari, MD, Principal Investigator — Gundersen Lutheran Health System
Locations (1):
- Gundersen Lutheran Health System, La Crosse, Wisconsin, United States

REFERENCES:
- [Background] Yang HL, Li ZZ, Sun YG. Reliability of ultrasonography in diagnosis of biliary lithiasis. Chin Med J (Engl). 1990 Aug;103(8):638-41. PMID 2122943
- [Background] Cronan JJ. US diagnosis of choledocholithiasis: a reappraisal. Radiology. 1986 Oct;161(1):133-4. doi: 10.1148/radiology.161.1.3532178.
- [Background] Shea JA, Berlin JA, Escarce JJ, Clarke JR, Kinosian BP, Cabana MD, Tsai WW, Horangic N, Malet PF, Schwartz JS, et al. Revised estimates of diagnostic test sensitivity and specificity in suspected biliary tract disease. Arch Intern Med. 1994 Nov 28;154(22):2573-81. PMID 7979854
- [Background] Einstein DM, Lapin SA, Ralls PW, Halls JM. The insensitivity of sonography in the detection of choledocholithiasis. AJR Am J Roentgenol. 1984 Apr;142(4):725-8. doi: 10.2214/ajr.142.4.725. PMID 6608231
- [Derived] Kothari SN, Obinwanne KM, Baker MT, Mathiason MA, Kallies KJ. A prospective, blinded comparison of laparoscopic ultrasound with transabdominal ultrasound for the detection of gallbladder pathology in morbidly obese patients. J Am Coll Surg. 2013 Jun;216(6):1057-62. doi: 10.1016/j.jamcollsurg.2013.02.009. Epub 2013 Apr 6. PMID 23571143

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasound Study Group
Started | 253
Completed | 253
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ultrasound Study Group
Number analyzed (Participants) | 253
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 251
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 43.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192
  Male | 61
Region of Enrollment [Number; unit: participants]
  United States | 253

OUTCOME MEASURES:

1. Primary Outcome: Cholelithiasis on Transabdominal Ultrasound Versus Laparoscopic Ultrasound.
Description: Number of patients with cholelithiasis.
Time Frame: transabdominal measurements within 30 days prior to surgery; laparoscopic ultrasound measurements are completed intraoperatively
Measure: Number; unit: participants
Groups:
- Transabdominal Ultrasound: Patients with no history of gallbladder surgery who are undergoing elective laparoscopic roux-en-Y gastric bypass that have consented to undergo a preoperative transabdominal ultrasound in addition to routine preoperative assessment for surgery.
- Laparoscopic Ultrasound: Laparoscopic ultrasound is performed intraoperatively at the time of gastric bypass.
Arm/Group | Transabdominal Ultrasound | Laparoscopic Ultrasound
Number analyzed (Participants) | 253 | 253
participants | 61 | 60
Statistical Analysis 1: Comparison: Transabdominal Ultrasound vs Laparoscopic Ultrasound; Test type: Superiority or Other; p = 0.763, Chi-squared

2. Secondary Outcome: Common Bile Duct (CBD) Diameter Measured by Transabdominal Ultrasound Versus Laparoscopic Ultrasound.
Description: Mean CBD diameter.
Time Frame: transabdominal measurements will be done within 30 days prior to surgery; laparoscopic ultrasound measurements are completed intraoperatively
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Laparoscopic Ultrasound: Laparoscopic ultrasound is performed intraoperatively during gastric bypass
Arm/Group | Transabdominal Ultrasound | Laparoscopic Ultrasound
Number analyzed (Participants) | 253 | 253
millimeters | 4.0 (1.28) | 3.7 (1.37)

3. Primary Outcome: Polyps on Transabdominal and Laparoscopic Ultrasound
Description: Number of patients with polyps.
Time Frame: 6 years
Measure: Number; unit: participants
Arm/Group | Transabdominal Ultrasound | Laparoscopic Ultrasound
Number analyzed (Participants) | 253 | 253
participants | 6 | 41
Statistical Analysis 1: Comparison: Transabdominal Ultrasound vs Laparoscopic Ultrasound; Test type: Superiority or Other; p < 0.001, Chi-squared

ADVERSE EVENTS:
Arm/Group | Ultrasound Study Group
Serious Adverse Events (participants affected / at risk) | 0/253
Other Adverse Events (participants affected / at risk) | 0/253

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes